CLINICAL TRIAL: NCT06495918
Title: A Phase 3, Multicenter, Double-Masked, Randomized, Parallel Group Study to Evaluate the Efficacy and Safety of Intravitreal OTX-TKI (Axitinib Implant) in Subjects With Neovascular Age- Related Macular Degeneration
Brief Title: Study to Evaluate the Efficacy and Safety of Intravitreal OTX-TKI (Axitinib Implant) in Subjects With Neovascular Age- Related Macular Degeneration
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Collaborators: Fortrea (Industry); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OTX-TKI-2023-AMD-303
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Neovascular Age-Related Macular Degeneration; Tyrosine Kinase Inhibitor; OTX-TKI
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- OTX-TKI Re-dose (Experimental)
  Interventions: Drug: OTX-TKI
- Aflibercept 2mg on label (Active Comparator)
  Interventions: Drug: Aflibercept
- Aflibercept 8mg high dose (Other)
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: OTX-TKI — Intravitreal Injection of OTX-TKI
  Arms: OTX-TKI Re-dose
Drug: Aflibercept — Intravitreal Injection of 2mg of aflibercept
  Arms: Aflibercept 2mg on label
Drug: Aflibercept — Intravitreal Injection of 8mg of aflibercept
  Arms: Aflibercept 8mg high dose

SUMMARY:
Study to Evaluate the Efficacy and Safety of Intravitreal OTX-TKI (Axitinib Implant) in Subjects with Neovascular Age- Related Macular Degeneration

ELIGIBILITY:
Inclusion Criteria:

* Treatment naïve juxtafoveal and/or SFNV secondary to Neovascular Age- Related Macular Degeneration (nAMD) with leakage involving the fovea in the study eye prior to Screening, or have a diagnosis of Neovascular Age- Related Macular Degeneration (nAMD) in study eye within 3 months prior to screening and received up to 2 monthly injections of 2 mg aflibercept with last injection approximately 4 weeks prior to Screening
* Have provided written consent

Exclusion Criteria:

* Monocular subject or Best Corrected Visual Acuity (BCVA) score of <20 ETDRS letters or 20/400 in fellow eye at Screening
* Have evidence of a scar, fibrosis, or atrophy of >50% of the total lesion in the study eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 825 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2027-01-08 (Estimated); Study Completion 2027-01-08 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) | Week 48
  Mean change in Best Corrected Visual Acuity (BCVA) from baseline at Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Dilsher Dhoot, MD, Principal Investigator — California Retina Consultants (CRC) - Santa Barbara
Locations (97):
- United States (84):
  - Associated Retina Consultant, Gilbert, Arizona
  - Associated Retina Consultants, Ltd., Phoenix, Arizona
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Retina Macula Institute of Arizona, Scottsdale, Arizona
  - California Retina Consultants, Bakersfield, California
  - The Retina Partners, Encino, California
  - Retina Consultants of Orange County, Fullerton, California
  - Atlantis Eyecare, Huntington Beach, California
  - Salehi Retina Institute, Inc., dba Retina Associates of Southern California, Huntington Beach, California
  - Kaiser Permanente Division of Research, Oakland, California
  - California Retina Consultants, Oxnard, California
  - Stanford Health Care - Byers Eye Institute, Palo Alto, California
  - Stanford University School of Medicine, Byers Eye Institute, Palo Alto, California
  - California Eye Specialists Medical Group, INC, Pasadena, California
  - Retinal Consultants Medical Group, Sacramento, California
  - Orange County Retina Medical Group, Santa Ana, California
  - California Retina Consultants, Santa Barbara, California
  - Macula Retina Vitreous Research Institute, Torrance, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Retina Consultants of Southern Colorado, Colorado Springs, Colorado
  - RSC Research, LLC, Denver, Colorado
  - Colorado Retina Associates, Lakewood, Colorado
  - Retina Consultants, P.C, Manchester, Connecticut
  - Retina Group of New England, Waterford, Connecticut
  - Advanced Research LLC., Deerfield Beach, Florida
  - Rand Eye Institute, Deerfield Beach, Florida
  - Retina Group of Florida, Fort Lauderdale, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - South Florida Retina Institute, Miami, Florida
  - Florida Retina Institude, Orlando, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - MedEye Associates, South Miami, Florida
  - Retina Vitreous Associates of Florida- Saint Petersburg, St. Petersburg, Florida
  - Retina Vitreous Associates of Florida, Tampa, Florida
  - Southeast Retina Center, Augusta, Georgia
  - University Retina and Macula Associates, PC, Oak Forest, Illinois
  - Illinois Retina Associates, Oak Park, Illinois
  - Springfield Clinic Opthalmology Department, Springfield, Illinois
  - Associate Vitreoretinal and Uveitis Consultants, Carmel, Indiana
  - Retina Partners Midwest, P.C., Carmel, Indiana
  - Retina Partners Midwest, Indianapolis, Indiana
  - Wolfe Clinic PC dba Wolfe Eye Clinic, West Des Moines, Iowa
  - The Retina Group of Washington - Chevy Chase, Chevy Chase, Maryland
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Mid Atlantic Retina Specialists, Hagerstown, Maryland
  - Retina Specialists - Towson Office, Towson, Maryland
  - Associated Retinal Consultants, P.C., Royal Oak, Michigan
  - Retina Consultants of Minnesota, Minneapolis, Minnesota
  - Mississippi Retina Associates, Madison, Mississippi
  - The Retina Institute, St Louis, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Envision Ocular, LLC, Bloomfield, New Jersey
  - Vision Research Center Eye Associates of New Mexico, Albuquerque, New Mexico
  - Retina Vitreous Surgeons of CNY, PC, Liverpool, New York
  - Asheville Eye Associates (AEA) - Asheville, Asheville, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - EyeHealth Northwest, Portland, Oregon
  - Erie Retina Research, Erie, Pennsylvania
  - Palmetto Retina Center, LLC, Aiken, South Carolina
  - Charleston Neuroscience Instititute, LLC, Beaufort, South Carolina
  - Palmetto Retina Center, LLC, Florence, South Carolina
  - Palmetto Retina Center, LLC, West Columbia, South Carolina
  - Black Hills Regional Eye Institute, LLP, Rapid City, South Dakota
  - Charles Retina Institute, Germantown, Tennessee
  - Southeastern Retina Associates PC, Johnson City, Tennessee
  - Tennessee Retina, PC, Nashville, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Texas Retina Associates, Arlington, Texas
  - Austin Research Center for Retina, Austin, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina Consultants of Texas, Beaumont, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Star Vision Research, Burleson, Texas
  - Texas Retina Associates, Dallas, Texas
  - Texas Retina Center, Houston, Texas
  - Retina Consultants of Texas, Katy, Texas
  - Retina Consultants of Texas, San Antonio, Texas
  - Retina Center of Texas, Southlake, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Retina Associates of Utah, Salt Lake City, Utah
  - Rocky Mountain Retina Consultants, Salt Lake City, Utah
  - Retina Group of Washington, Fairfax, Virginia
  - Vistar Eye Center, Roanoke, Virginia
  - Eye Clinic of Wisconsin, SC, Wausau, Wisconsin
- Argentina (10):
  - Organización Médica de Investigación (OMI), Buenos Aires
  - Centro Privado de Ojos, Buenos Aires
  - Charles Research Center (Centro Oftalmologico Dr. Charles S.A), Buenos Aires
  - Buenos Aires Macula, Caba
  - Instituto Oftalmologico de Buenos Aires SA - OFTALMOS, Caba
  - Fundacion Zambrano - Cirugia Ocular, Caba
  - Fundacion Jorge Zambrano para la investigacion, Diagnostico y Tratamiento de las enfermedades oculares, Ciudad Autonoma de Buenos Aire
  - Oftar Mendoza Srl Centro Privado de Oftalmologia, Mendoza
  - Centro Vision S.A., Mendoza
  - Laser Vision Group, Rosario
- Australia (2):
  - Albury Eye Clinic, Albury, New South Wales
  - Marsden Eye Specialists (MES) - Parramatta, Parramatta, New South Wales
- Emanuelli Research and Development Center, LLC, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: No